CLINICAL TRIAL: NCT04784520
Title: A Multicentre, Open-label, Single-arm Phase II Study of HA121-28 Tablets in Advanced Biliary Tract Cancer (BTC)
Brief Title: A Study of HA121-28 Tablets in Advanced Biliary Tract Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The primary endpoint did not meet expectation.
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HA122-CSP-002
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HA121-28 tablets (Experimental): HA121-28 600 mg, po, QD×21 days, every 4 weeks (28 days)
  Interventions: Drug: HA121-28 tablets

INTERVENTIONS:
Drug: HA121-28 tablets — HA121-28 600 mg, po, QD×21 days, every 4 weeks (28 days)

SUMMARY:
This study is a multicenter, open-label, single-arm phase II study to evaluate efficacy, safety, and pharmacokinetics characteristics of HA121-28 tablets in advanced biliary tract cancer (BTC). A total of approximately 30 subjects with advanced BTC will be enrolled. The subjects will undergo a 3 weeks-on and 1week-off treatment scheme with HA121-28 tablets 600 mg orally once daily in the 28-day cycle until disease progression or intolerable toxic reaction, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Be willing to participate in the clinical trial and sign the informed consent;
* Histologically/cytologically confirmed unresectable locally advanced or metastatic BTC (including cholangiocarcinoma or gallbladder cancer) with failure of or intolerance to the prior therapy (including disease progression within 6 months after adjuvant chemotherapy) and with at least one measurable lesion based on RECIST 1.1 criteria;
* Aged 18 to 75 years (inclusive);
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0~1;
* Routine blood test results must meet the following criteria without blood transfusion within 14 days: 1) Hemoglobin (Hb)≥90 g/L; 2) Absolute neutrophil count (ANC)≥1.5 x 10^9/L; 3) Platelet count (PLT)≥75×10^9/L;
* Coagulation test results must meet the following criteria: International Normalized Ratio (INR) <1.5 or Activated Partial Thromboplastin Time (APTT) <1.5×ULN;
* Other laboratory test results must meet all the following criteria: 1) Total bilirubin (TBIL)≤1.5×ULN, Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤2.5×ULN (TBIL≤3×ULN, ALT and AST≤5×ULN in the subjects with liver metastasis); 2) Serum creatinine≤1.5×ULN；3) Serum albumin≥28g/L;
* Male and female subjects of childbearing potential must agree to take effective contraception for the duration of treatment and for 6 months after completion of study drug administration; female subjects must have negative results of serum/urine pregnancy test within 7 days prior to enrollment and must not be breastfeeding.

Exclusion Criteria:

* Subjects with ampullary carcinoma;
* Subjects who had participated in other clinical trials and received the treatment within 4 weeks prior to enrolment;
* The time interval between the end of the last antitumor treatment and the first administration of HA121-28 tablets < 4 weeks (for any antitumor treatment, including but not limited to chemotherapy, radiotherapy and targeted therapy), or < 2 weeks (for local palliative radiotherapy for pain relief or traditional Chinese medicine with approved indications for cancer);
* Urine protein≥2+ and urine protein > 1.0g/24h;
* History of other malignancies within the past 5 years prior to enrolment, except for cured cervical carcinoma in situ, non-melanoma skin cancer, superficial bladder tumor, and early esophageal and gastrointestinal cancers that were confined to the mucosal layer and resected under endoscopy;
* History of any solid-organ or bone-marrow transplantation (except the transplantation without immunosuppression such as corneal and hair transplantation);
* Unremitted toxic reaction>grade 1 due to any previous treatment at the time of enrollment (except for hair loss and pigmentation) which is considered to influence the safety evaluation;
* ECG meets one of the following criteria: 1) QT/QTc interval≥450ms, congenital long QT syndrome (LQTS) or family history of LQTS; 2) any clinically significant abnormalities of rhythm, conduction or morphology in the resting ECG requiring therapeutic intervention;
* Left ventricular ejection fraction (LVEF) <50% in echocardiogram;
* Severe concomitant diseases which may have influence on the safety of the subjects or the completion of the study based on the investigator' judgement such as uncontrolled hypertension (systolic pressure ≥150 mmHg or diastolic pressure ≥100 mmHg after treatment);
* High risk factors of gastrointestinal diseases such as gastrointestinal perforation and abdominal fistula;
* Subjects with spinal cord, meningeal or brain metastasis (except for asymptomatic or stable brain metastasis within 4 weeks prior to administration);
* Subjects with hepatopathy meet one of the following criteria: 1) HBsAg positive and HBV DNA >2000 IU/mL（or >1×10^4 copies/mL）; 2) HCV antibody positive and HCV RNA positive; 3) cirrhosis;
* HIV antibody positive;
* Subjects have history of surgery within 4 weeks prior to administration or have not been recovered from any previous invasive procedure, except for biliary stenting, biliary drainage, etc.;
* Not suitable for the study in the investigator's opinion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
progression-free survival | Approximately 3.5 years

SECONDARY OUTCOMES:
objective remission rate | Approximately 3.5 years
overall survival | Approximately 3.5 years
disease control rate | Approximately 3.5 years
duration of response | Approximately 3.5 years

OTHER OUTCOMES:
adverse events incidence | Approximately 3.5 years
HA121-28 plasma concentration | Approximately 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - The First Affiliated Hospital，Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guanzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No